CLINICAL TRIAL: NCT00760357
Title: A Retrospective Analysis of Patients With Full Thickness Wounds in Limbs With Critical Ischemia
Status: Completed | Type: Observational
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Principal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-007
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Critical Limb Ischemia
Keywords: Critical Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Once the patients are identified that have a full thickness wound on a limb clearly identified as having critical limb ischemia, these patients will be evaluated. The data that will be extracted from each chart will include patient's age, patient's gender, number of office visits, presence of diabetes, presence of osteomyelitis, type and amount of antibiotic administered, number of hyperbaric oxygen treatments, and if the wound healed.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Retrospective Anaylsis: Once the patients are identified that have a full thickness wound on a limb clearly identified as having critical limb ischemia, these patients will be evaluated

SUMMARY:
Once the patients are identified that have a full thickness wound on a limb clearly identified as having critical limb ischemia, these patients will be evaluated. The data that will be extracted from each chart will include patient's age, patient's gender, number of office visits, presence of diabetes, presence of osteomyelitis, type and amount of antibiotic administered, number of hyperbaric oxygen treatments, and if the wound healed.

DETAILED DESCRIPTION:
Clinicians have even learned to group patients into different etiologic categories based on underlying disease such as diabetes mellitus, decubitus ulcer, surgical site infection, venous insufficiency, arterial insufficiency and others. It seems that wounds have been grouped into these categories because of their common barriers, which should allow us more precise algorithms and may provide better outcomes. That is diabetics tend to have the barriers of poor perfusion, endothelial cell dysfunction, white blood cell dysfunction, hyperglycemia, neuropathy and repetitive trauma. Venous insufficiency patients tend to have perivascular cuffing and peri wound edema. However patients with venous leg ulcers commonly have peripheral arterial disease and diabetes (3). The point is regardless of the etiology of the wound every patient must be evaluated for all barriers on every visit. Arbitrarily dividing chronic wounds in the etiologic categories has not significantly improved wound healing outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the study are patients that demonstrate the following:

  * A limb with a TCpO2 less than 20 with a full thickness wound.
  * Initial visit from August 1, 2002 to December 31, 2005.

Exclusion Criteria:

* The exclusion criteria for the study are patients that demonstrate the following:

  * Partial thickness wound or no wound in limb with critical ischemia.
  * A medical record that does not clearly demonstrate critical limb ischemia or does not clearly demonstrates a full thickness wound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Once the patients are identified that have a full thickness wound on a limb clearly identified as having critical limb ischemia, these patients will be evaluated. The data that will be extracted from each chart will include patient's age, patient's gender, number of office visits, presence of diabetes, presence of osteomyelitis, type and amount of antibiotic administered, number of hyperbaric oxygen treatments, and if the wound healed.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Once the patients are identified that have a full thickness wound on a limb clearly identified as having critical limb ischemia, these patients will be evaluated | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Randall D Wolcott, MD, Principal Investigator — Southwest Regional Wound Care Center
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States